CLINICAL TRIAL: NCT05182697
Title: A Randomized, Double-Blind, Sparing-effect Placebo Controlled, With Cross-over Study to Evaluate the Safety, Tolerability and Efficacy of SCI-210 in Children With Autism Spectrum Disorder (ASD)
Brief Title: SCI-210 in the Treatment of Children and Young Adults With AutismEvaluate the Safety, Tolerability and Efficacy of SCI-210 in Children With Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurothera Labs Inc. (Industry)
Collaborators: Negev Autism Center Soroka University Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCRC21013
Record Dates: First submitted 2021-11-29; First posted 2022-01-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCI-210 (Experimental): Oral CBD oil plus pills of CannAmide (palmitoylethanolamide (PEA) 400 mg twice daily
  Interventions: Drug: SCI-210
- CBD oil (Active Comparator): CBD- active CBD oil with twice daily and CannAmide Placebo pills matched in appearance and taste to CannAmide active pill.
  Interventions: Drug: Oral CBD oil

INTERVENTIONS:
Drug: SCI-210 — Oral CBD oil plus pills of CannAmide (palmitoylethanolamide (PEA) 400 mg twice daily
  Arms: SCI-210
Drug: Oral CBD oil — CBD- active CBD oil with twice daily CannAmide Placebo pills matched in appearance and taste to CannAmide active pill.
  Arms: CBD oil

SUMMARY:
To evaluate the safety and efficacy of SCI-210 in the treatment of Autism Spectrum Disorders (ASD)

DETAILED DESCRIPTION:
The innovative compound SCI-210 consists of CBD oil combined with CannAmide (PEA formulation) using the "entourage effect" to enhance efficacy of CBD. It is believed that PEA potentiates anandamide responses in non-vascular tissues. This effect is called "entourage effect". The "entourage effect" can be achieved by enhancing the action of endogenous anandamide through an increase in the affinity for receptors and/or a decrease in enzymatic degradation of anandamide (primarily by fatty acid amide hydrolase, FAAH). Thus, the combination of CBD oil with PEA is believed to be more effective than CBD oil alone, while AEs are not increased by the addition of the natural substance PEA.

SCI-210 has not been tested in clinical trials before, but anecdotal evidence of combined use of CBD and CannAmide in ASD patients has been accumulated in recent months. The evidence suggests the beneficial effects of the combination in alleviating ASD symptoms with no reported adverse events associated with the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged between 5 and 18 years of age (inclusive)
2. Diagnosis of ASD confirmed by the ADOS-2 and DSM-5 criteria
3. Moderate or greater behavioral problems as measured by a rating of moderate or higher (≥4) on the Clinical Global Impression-Severity (CGI-S)
4. Presence of a parent/legal guardian who is able to consent for their participation and completes assessments regarding the child's development and behavior throughout the study
5. Patients eligible for cannabis treatment as regulated by the Israeli Ministry of Health, as out lined in the Medical Cannabis unit circular on Licenses for cannabis use, Procedure number 106, version 5 dated Jan 2021

Exclusion Criteria:

1. Children who are already receiving cannabis, antipsychotic drugs, or stimulants.
2. Children with heart, liver, renal or hematological disorders.
3. History of active seizure disorder or epilepsy; patients who are seizure free for more than 3 years can take part in the study
4. Exposure to any investigational agent in the 30 days prior to trial onset.
5. A current psychiatric diagnosis of bipolar disorder, major depressive disorder (MDD), psychosis, schizophrenia, or post-traumatic stress disorder (PTSD)
6. Subjects who have had changes in non-exclusionary psychotropic medications within 4 weeks of initiation of trial.
7. Allergic to cannabinoids or PEA tablet components.
8. History of substance abuse (including alcohol abuse or dependence) or laboratory evidence of drug abuse on the Visit 1 drug-screening panel.
9. Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he or she were to participate in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety of SCI-210 in the treatment of Autism Spectrum Disorders (ASD) | 24 weeks
  Evaluation of the safety of SCI-210 in the treatment of Autism Spectrum Disorders (ASD) throughout the 24 week treatment period.
  Adverse effects will be assessed using an adverse effects checklist (AEC) containing 19 items from the Liverpool Adverse Events Profile (LAEP) in addition to 15 items that have been used previously to assess side effects of CBD. These will be compared between the groups. Dropout rates from study will also be compared between these groups.
Evaluation of the efficacy of SCI-210 in the treatment of Autism Spectrum Disorders (ASD) | 24 weeks
  Evaluation of the efficacy of SCI-210 in the treatment of Autism Spectrum Disorders (ASD) throughout the 24 week treatment period.
  The primary outcome measures of the study will be the Clinical Global Impressions-Improvement (CGI-I) performed by a clinician. These will be completed at the beginning (Time 0), middle (4 weeks) and end (8 weeks) of each stage. Efficacy of treatment will be evaluated by comparing the change in CGI-I scores during the different periods of the study between the two treatment and control groups.
Evaluation of the efficacy of SCI-210 in the treatment of Autism Spectrum Disorders (ASD) | 24 weeks
  Evaluation of the efficacy of SCI-210 in the treatment of Autism Spectrum Disorders (ASD) throughout the 24 week treatment period.
  The primary outcome measures of the study will be the Aberrant Behavior Checklist-Community (ABC-C) parent questionnaire performed by a clinician. These will be completed at the beginning (Time 0), middle (4 weeks) and end (8 weeks) of each stage. Efficacy of treatment will be evaluated by comparing the change in ABC-C scores during the different periods of the study between the two treatment and control groups.

SECONDARY OUTCOMES:
Evaluate the safety of SCI-210 in children with ASD. | 24 weeks
  Evaluate the safety of SCI-210 in children with ASD throughout the 24 week treatment periodAdverse effects will be assessed using an adverse effects checklist (AEC) containing 19 items from the Liverpool Adverse Events Profile (LAEP) in addition to 15 items that have been used previously to assess side effects of CBD. These will be compared between the groups. Dropout rates from study will also be compared between these groups.
Evaluate the tolerability of SCI-210 in children with ASD. | 24 weeks
  Evaluate the tolerability of SCI-210 in children with ASD throughout the 24 week treatment period Adverse effects will be assessed using an adverse effects checklist (AEC) containing 19 items from the Liverpool Adverse Events Profile (LAEP) in addition to 15 items that have been used previously to assess side effects of CBD. These will be compared between the groups. Dropout rates from study will also be compared between these groups.
Assess the efficacy of SCI-210 in reducing disruptive behaviors among children with ASD | 20 weeks
  Parents will fill out the following questionnaire at the beginning (Time 0) of the trial and at the end of the first (8 weeks) and second (20 weeks) stage:
  The Social Responsiveness Scale (SRS) will be used to estimate changes in the social abilities of the child.
  A total composite score between 60 and 65 is associated with mild to moderate deficits in social interaction. Scores between 66 and 75 are considered to display a moderate deficit in social interaction, and a score greater than 76 is considered severe and strongly associated with the clinical diagnosis of ASD
Assess the efficacy of SCI-210 in reducing sleep problems among children with ASD | 20 weeks
  Parents will fill out the following questionnaire at the beginning (Time 0) of the trial and at the end of the first (8 weeks) and second (20 weeks) stage:
  The Children's Sleep Habit Questionnaire (CSHQ) will be used to estimate changes in the sleep quality of the child.
  A Total Sleep Disturbances score is calculated as the sum of all CSHQ scored questions, and can range from 33 to 99. A Total Sleep Disturbances score of over 41 indicates a pediatric sleep disorde.
Assess the efficacy of SCI-210 in reducing ASD symptoms among children with ASD. | 20 weeks
  Children will participate in the following assessment at the beginning (Time 0) of the trial and at the end of the first (8 weeks) and second (20 weeks) stage:
  The Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2) will be used to estimate changes in core ASD symptoms.
  The comparison score ranges from 1-10, where 1 indicates minimal-to-no evidence of autism-related symptoms and 10 indicates a high level of impairment.
Assess the efficacy of SCI-210 in improving adaptive behaviors among children with ASD | 20 weeks
  Parents will fill out the following questionnaire at the beginning (Time 0) of the trial and at the end of the first (8 weeks) and second (20 weeks) stage:
  The Adaptive Behavior Assessment System 3rd edition (ABAS-3) will be used to estimate changes in the adaptive behaviors of the child.
  The ratings given for each skill area are converted into a score from 1 to 19, with 1 being the lowest and 19 being the highest, and scores of 8 to 12 being in the Average range
Assess the efficacy of SCI-210 in improving language abilities among children with ASD | 20 weeks
  Children will participate in the following assessment at the beginning (Time 0) of the trial and at the end of the first (8 weeks) and second (20 weeks) stage:
  The Preschool Language Scale will be used to estimate changes in language abilities.
  A standard score of 100 on this scale represents the performance of the typical student of a given age. Standard scores between 85 and 115 correspond to one standard deviation below and above the mean, respectively; scores within this range are considered to be within normal limits.
Assess the effects of SCI-210 on eye tracking measures when viewing social movies. | 20 weeks
  Eye tracking assessment will be performedat the beginning (Time 0) of the trial and at the end of the first (8 weeks) and second (20 weeks) stage Eye tracking while watching movies will be performed to estimate changes in the way the children observe movies with social information (e.g., children playing). This will quantify changes in the social preferences of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Gal Meiri, MD, MHA, Principal Investigator — Clinical Research Center and Negev Autism Center Soroka University Medical Center, Be'er-Sheva, Israel
Locations (1):
- Clinical Research Center and Negev Autism Center Soroka University Medical Center, Be'er-Sheva, Israel, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No